CLINICAL TRIAL: NCT03037866
Title: Primary Prevention of Sexual Violence Among College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Health Promotion Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Kenneth W Griffin, Senior Research Scientist, National Health Promotion Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44DA039602-01 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-31 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Sexual Violence; Substance Use; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LifeSkills Training for College (Experimental): All students who consent to participate in the proposed study will complete pre, post, six- and 12-month follow-up surveys. Those randomized to the intervention group (n=2000) will participate in the LST program adapted for college which consists of six 30-minute online sessions (content-specific instruction and skills building activities along with opportunities to apply newly acquired knowledge and practice new skills) and three 60-minute small groups sessions (facilitator-led sessions with fellow incoming students that complement the online modules).
  Interventions: Behavioral: LifeSkills Training for College
- Treatment as Usual (Control) (No Intervention): All students who consent to participate in the proposed study will complete pre, post, six- and 12-month follow-up surveys. Those randomized to the control group (n=2000) will not participate in LST but will receive the sexual violence and substance abuse educational content normally provided by their schools.

INTERVENTIONS:
Behavioral: LifeSkills Training for College — The intervention will consist of e-learning modules (self-guided) and small-group sessions (facilitator led). The intervention is designed for new college students and is aimed at providing tools and strategies to help them maximize opportunities and adeptly handle the challenges ahead. The intervention will teach them the knowledge and skills needed to stay safe from problems that are prevalent among new students on college campuses, such as alcohol and drug abuse and sexual violence.
  Other Names: LifeSkills Training; LST
  Arms: LifeSkills Training for College

SUMMARY:
This project is designed to address the urgent need for an effective primary prevention approach to the problem of sexual violence among college students. The project involves developing, feasibility testing, and testing for effectiveness an innovative new approach to the primary prevention of sexual violence, alcohol, and drug abuse among college students utilizing both online e-learning and small group facilitator-led intervention modalities. The intervention is an adaptation of the successful evidence-based substance abuse and violence prevention approach called Life Skills Training (LST). The adapted intervention is designed to address the relationship between sexual violence and substance abuse; positively change social norms surrounding alcohol/drug abuse and sexual violence; train bystanders to identify and appropriately respond to problematic situations; and build social, self-regulation, and relationship skills through interactive learning and behavioral rehearsal scenarios. At the conclusion of the study, the investigators expect to be able to widely disseminate and market a new evidence-based primary prevention intervention for sexual violence for use in a variety of higher educational settings.

DETAILED DESCRIPTION:
This proposal is designed to address the urgent need for an effective primary prevention approach to the problem of sexual violence among college students. It is estimated that 1 in every 5 college women has been sexually assaulted while in college. There is a dearth of primary prevention strategies that have demonstrated significant reductions in sexual violence in college students as part of a rigorously designed evaluation. Research shows that many victims of sexual assault are abused while drunk, under the influence of drugs, or otherwise incapacitated, and that incidents of sexual violence typically occur in college party settings where the victim knows the perpetrator and the perpetrator has been drinking or using drugs. In Phase I of this study, the investigators established the feasibility, relevance, and appeal of the new primary prevention program for sexual violence, alcohol, and drug abuse for incoming college students. The program is an adaptation of a successful evidence-based substance abuse and violence prevention approach called Life Skills Training (LST). The LST approach is designed to build personal self-management skills, social skills, and other life skills needed to reduce substance abuse and violence, increase resilience, and successfully navigate developmental tasks. In Phase I, the investigators developed the full scope and sequence of the program which outlines the learning objectives and activities of the of the online e-learning modules and small group facilitator-led sessions; developed relevant prototype materials to represent a subset of the full program; conducted formative research to establish the feasibility, relevance, and appeal of the intervention through a series of focus groups with college students and key informant interviews with college prevention staff; and recruited over 40 colleges and universities to participate in Phase II of the project. In Phase II, the investigators will fully develop the skills building curriculum materials and conduct a rigorous randomized controlled trial to examine the impact of the intervention. Forty colleges will be randomized into either an intervention group that will receive the new intervention or a treatment-as-usual control group that will receive the existing information on sexual violence provided at the school. At the end of a two-month intervention period, and at 6- and 12month follow-up assessments, the investigators will compare changes in behaviors, norms, attitudes, and knowledge regarding alcohol, drug abuse, and sexual violence. The ultimate intervention holds promise for wide dissemination as an evidence-based primary prevention approach for sexual violence to four-year colleges, community or junior colleges, universities, graduate and professional schools, for-profit schools, trade schools, and career and technical schools.

Phase II Specific Aims

1. Fully develop the sexual violence primary prevention skills building curriculum materials;
2. Conduct a randomized controlled trial to examine the impact of the intervention; randomize 40 colleges into either an intervention group that will receive the new intervention or a treatment-as-usual control group that will receive the existing information on sexual violence provided at the school;
3. Conduct an outcome evaluation by assessing changes in the two experimental conditions with regards to behaviors, norms, attitudes, and knowledge regarding alcohol, drug abuse, and sexual violence at the end of the two-month intervention period, and at 6- and 12-month follow-up assessments;
4. Conduct a process evaluation to document and monitor all Phase II project activities;
5. Disseminate research findings to the scientific and practice communities;
6. Create a provider training mechanism to promote dissemination and sustainability of the intervention;
7. Based on the commercialization plan, implement a marketing strategy for the new primary prevention program aimed at institutions of higher education across the country.

ELIGIBILITY:
Inclusion Criteria:

* College students

Exclusion Criteria:

* Significant cognitive impairment or severe learning disabilities, as screened by field staff at participating sites
* Any previous experience with the intervention program will also exclude adolescents from participating

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4000 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Sexual violence behaviors, norms, and attitudes at baseline | Pre-test (prior to participating in the first session/module of the intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding sexual violence and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline sexual violence behaviors, norms, and attitudes at post-intervention | Post-test (within 2 weeks of completing final session/module of the intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding sexual violence and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline sexual violence behaviors, norms, and attitudes at 6-months | 6-month followup (within 6-7 months of completing final session of intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding sexual violence and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline sexual violence behaviors, norms, and attitudes at 12-months | 12-month followup (within 12-13 months of completing final session of intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding sexual violence and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.

SECONDARY OUTCOMES:
Substance use and abuse behaviors, norms, and attitudes at baseline | Pre-test (prior to participating in the first session/module of the intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding alcohol and drug abuse and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline substance use and abuse behaviors, norms, and attitudes at post-intervention | Post-test (within 2 weeks of completing final session/module of the intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding alcohol and drug abuse and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline substance use and abuse behaviors, norms, and attitudes at 6-months | 6-month followup (within 6-7 months of completing final session of intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding alcohol and drug abuse and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Change in baseline substance use and abuse behaviors, norms, and attitudes at 12-months | 12-month followup (within 12-13 months of completing final session of intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding alcohol and drug abuse and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Griffin, PhD, Principal Investigator — National Health Promotion Associates, Inc.

IPD SHARING:
Plan to Share IPD: No